CLINICAL TRIAL: NCT00997087
Title: Phase IIa A Randomized, Double-Blind, Placebo-Controlled Trial of Flumazenil for the Treatment of Obsessive Compulsive Disorder.
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Flumazenil for the Treatment of Obsessive Compulsive Disorder
Acronym: OCD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study completed and data was inconclusive.
Sponsor: Parkway Medical Center (Other)
Responsible Party: Principal Investigator, James G.Sullivan, MD, Principal Investigator, Parkway Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JGS-001
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Flumazenil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill, Placebo (Placebo Comparator)
  Interventions: Drug: Flumazenil
- Flumazenil (Active Comparator)
  Interventions: Drug: Flumazenil

INTERVENTIONS:
Drug: Flumazenil — Sublingual daily

SUMMARY:
The purpose of this study is to evaluate the efficacy of flumazenil in the outpatient treatment of Obsessive Compulsive Disorder (OCD).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide written informed consent.
* Age 19-60, inclusive.
* Diagnosis documented according to DSM-IV of OCD.
* Exhibits moderate to severe OCD symptoms and a minimum score of 16 or greater -YBOCS at screening.
* Willing and able to discontinue current medications taken for the treatment of OCD.
* Able to attend and participate in all study visits.
* Agree to continue if in current psychosocial therapy throughout the remainder of the study.
* If female and of child-bearing potential, willing to use an acceptable method of birth control for the duration of the study.
* If male, willing to use barrier method of birth control or had previous vasectomy.

Exclusion Criteria:

* Have other DSM-IV Axis I diagnoses.
* Pregnant as confirmed by urine analysis, or lactating, or unwilling to comply with use of contraception.
* Unwilling or unable to washout (discontinue) from prohibited medications such as antidepressants (See Appendix 2).
* Depression symptoms with a score of 15 or greater on the MADRS at screening.
* Current suicidal ideation or plan within the last 30 days.
* Have a medical condition which, in the opinion of the investigator, makes study participation unsafe or noncompliant.
* Abnormal physical exam or laboratory values which, in the opinion of the investigator, makes study participation unsafe or may require introduction of concomitant medications during the course of the study.
* Benzodiazepine and/or similar sedative-hypnotic or anxiolytic use or abuse within 15 days of potential flumazenil treatment: patients must not be habituated to benzodiazepines and must provide a urine sample that is negative for benzodiazepines, must not be taking supra-therapeutic doses of zolpidem (AmbienTM) or zaleplon (SonataTM ). (See Appendix 2).
* Patients who are taking Phenobarbital for a documented seizure disorder can be admitted. Patients with a seizure disorder being managed with clonazepam (KlonopinTM ) or other benzodiazepine cannot participate, patients must not be taking TCA, lithium, methylxanthines, isoniazid, propoxyphene, monoamine oxidase inhibitors, bupropion HCL, and cyclosporine. (See Appendix 2).
* Previously treated with flumazenil for OCD.
* AIDS as determined by self-report.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Score | 12 weeks

SECONDARY OUTCOMES:
Safety will be assessed by Adverse Events, Changes in physical exam, laboratory values. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James G Sullivan, MD, Principal Investigator — Parkway Medical Center
Locations (1):
- James G. Sullivan, MD, Birmingham, Alabama, United States